CLINICAL TRIAL: NCT04961073
Title: The Prevalence of Multiple Risk Behaviours and Its Association With Health Consequence Among Hong Kong Chinese Adults
Brief Title: Prevalence of Multiple Risk Behaviours and Its Association With Health Consequence
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: NCD survey UW 21-440
Record Dates: First submitted 2021-06-19; First posted 2021-07-14 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-07

CONDITIONS: Non-communicable Diseases
Keywords: Risk behaviours; Health consequence; Non-communicable diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hong Kong is facing an increasing threat of non-communicable diseases (NCDs), which is compounded by population aging. In 2016, 25,771 registered deaths (approximately 55%) were attributed to NCDs. In addition, NCDs caused 104,600 potential years of life lost before 70 years of age. WHO has identified four major behavioral risk factors - tobacco use, harmful use of alcohol, an unhealthy diet, and physical inactivity - that contribute substantially to NCDs and can increase the risk of death. Most premature deaths from NCDs are preventable via lifestyle modification. Therefore, helping people adopting healthy lifestyle practices, such as having a balanced diet and engaging in irregular physical activity, and quitting health-risk behaviors, such as smoking and harmful use of alcohol can help prevent NCDs and improve the quality of life and overall health of the population. However, many people are unmotivated or find it difficult to modify their risk behaviors, despite their awareness of the associated health hazards.

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs), including cardiovascular diseases, cancers, diabetes and chronic respiratory diseases, are the most common and preventable causes of morbidity and mortality both globally and locally. According to the World Health Organization (WHO), 41 million (71%) of the 57.7 million global deaths each year are attributed to NCDs. NCDs are often associated with older age groups, but evidence shows that more than 15 million of all deaths attributed to NCDs occur between the ages of 30 and 69 years. The total number of annual deaths of NCDs will further increase to 55 million by 2030 unless urgent preventive measures are taken.

Hong Kong is facing an increasing threat of NCDs, which is compounded by population ageing. In 2016, 25,771 registered deaths (approximately 55%) were attributed to NCDs. In addition, NCDs caused 104,600 potential years of life lost before 70 years of age.

WHO has identified four major behavioural risk factors - tobacco use, harmful use of alcohol, an unhealthy diet and physical inactivity - that contribute substantially to NCDs and can increase the risk of death. Most premature deaths from NCDs are preventable via lifestyle modification. Therefore, helping people adopting healthy lifestyle practices, such as having a balanced diet and engaging in regular physical activity, and quitting health-risk behaviours, such as smoking and harmful use of alcohol can help prevent NCDs and improve quality of life and the overall health of the population. However, many people are unmotivated or find it difficult to modify their risk behaviours, despite their awareness of the associated health hazards. Our previous studies showed that many smokers continued to smoke even after receiving a diagnosis of cancer, diabetes or cardiovascular disease. In addition, health risk behaviours co-occur in clusters and that many people exhibit multiple risk behaviours. A sample of 16,818 adults from the 1998 US National Health Interview Survey revealed that 52% had two or more risk behaviours, including physical inactivity, overweight, cigarette smoking and risky drinking. Our previous study in Hong Kong also found associations between smoking and physical inactivity, an unhealthy diet and alcohol consumption. People with multiple health risk behaviours are usually associated with a higher increased risk of NCDs and face more challenges in the adoption of a healthy lifestyle than those with a single health risk behaviour. A review of the literature reveals that most interventions have been developed and evaluated targeted at people with single risk behaviour rather than multiple risk behaviours. It is crucial therefore to develop and evaluate appropriate interventions that targeting people with multiple risk behaviours with the aim to help them quit health-risk behaviours and adopt a healthy lifestyle, either sequentially or concurrently. First, however, a thorough understanding of the clustering of multiple health risk behaviours and the factors associated with such behaviours are crucial before any appropriate interventions can be developed and evaluated. The aim of the study is to investigate the prevalence of multiple risk behaviours and their association with health consequences among people aged 30 years or above. The objectives of the study are:

1. To investigate the clustering patterns of multiple health risk behaviours;
2. To identify factors associated with multiple risk behaviours; and
3. To find out the association between risk behaviours and non-communicable diseases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 years or above
* Able to speak Cantonese

Exclusion Criteria:

* Unable to speak Cantonese

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A randomized sample of Hong Kong Chinese adults who aged 30 years or above will be recruited at hotspots in eighteen districts in Hong Kong.
Sampling Method: Probability Sample
Enrollment: 5737 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Demographic data questionnaire | Baseline
  Personal demographic characteristics (e.g. sex, age, educational attainment, marital status, occupation, household income)
History of NCDs questionnaire | Baseline
  NCDs characteristics
Medical check-up questionnaire | Baseline
  History of medical check-up
Diet habits questionnaire | Baseline
  Personal habits of diet (e.g. daily vegetable and fruit intake)
Physical activity questionnaire | Baseline
  Personal habits of diet and physical activity (e.g. daily physical activity amount and time)
Unhealthy behaviors questionnaire | Baseline
  Habits of risky behaviors (e.g. smoking/ alcohol habits, daily cigarette consumption)
Knowledge and awareness of COVID-19 and NCDs questionnaire | Baseline
  Knowledge and awareness of COVID-19 and NCDs (e.g. knowledge about relationship between smoking and COVID, relationship between NCDs and COVID, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — School of Nursing, the University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project has been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)